CLINICAL TRIAL: NCT03182933
Title: Impact of Liposomal Bupivacaine Injected for Adductor Canal Block on Recovery Profile and Block Characteristics Following Total Knee Arthroplasty.
Brief Title: Liposomal Bupivacaine Versus Standard Bupivacaine in the Adductor Canal for Total Knee Arthroplasty
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated due to surgeon preferences
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-0869
Record Dates: First submitted 2017-06-01; First posted 2017-06-09 (Actual); Results first posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Pain
Keywords: 10 meter walk test; Opioid consumption
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liposomal bupivacaine group (Experimental): 20ml 1.33% liposomal bupivacaine administered in adductor canal (a type of peripheral nerve block)
  Interventions: Drug: Peripheral Nerve Blockade; Behavioral: 10 meter walk test on post-operative day 1; Other: In person and over the phone questionnaire; Device: Force transduction of quadriceps strength
- Standard bupivacaine group (Active Comparator): 20ml 0.5% standard bupivacaine in adductor canal (a type of peripheral nerve block)
  Interventions: Drug: Peripheral Nerve Blockade; Behavioral: 10 meter walk test on post-operative day 1; Other: In person and over the phone questionnaire; Device: Force transduction of quadriceps strength

INTERVENTIONS:
Drug: Peripheral Nerve Blockade — Each study arm will receive their respective formulation of local anesthetic, either standard bupivacaine or liposomal bupivacaine upon randomization
Behavioral: 10 meter walk test on post-operative day 1 — Patient asked to walk 10 meters at comfortable pace on post-operative day one when deemed safe to do so by the physical therapist
Other: In person and over the phone questionnaire — Presuming the patient has left the hospital each patient will be called on post-operative day 2, 3 to assess nausea, opioid consumption, satisfaction with anesthesia technique, nausea and vomiting as well as pain scores
Device: Force transduction of quadriceps strength — Patient will be asked to flex quadriceps at maximal ability and a transducer (Kiio device) will record a force value pre operatively and on post operative day 1

SUMMARY:
Study will evaluate the effect of liposomal bupivacaine versus standard bupivacaine on physical therapy measures and pain scores as well as opiate consumption.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) can be associated with a large amount of postoperative pain. This pain can oftentimes be severe enough to limit participation in physical therapy and ultimately delay discharge resulting in increased cost. Several strategies have been developed in an effort to decrease postoperative pain following TKA while maintaining lower extremity strength and maximizing participation in physical therapy. Recently, adductor canal blockade has gained popularity as it is reported to provide analgesia to the anterior knee without resulting in significant quadriceps muscle weakness. One downside of single shot peripheral blockade is the duration of analgesia can oftentimes be short lived. The advent of depot local anesthetics has made this an attractive option, especially in busy practices where placing peri-neural catheters may not be practical or cost effective. This study aims to carefully evaluate this relationship using a physical therapy evaluation method that relies on both motor strength and pain control. In addition, we hope to carefully evaluate motor strength using a novel method of strength measurement in an effort to further evaluate the impact of depot local anesthetic injection into the adductor canal on physical therapy and analgesia.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is scheduled for elective unilateral TKA;
2. The subject is ≥ 18 years and ≤ 80 years;
3. The subject's weight is between 65-130 kg;
4. The subject's primary anesthesia care team has planned for a neuraxial anesthetic (i.e. spinal, epidural or combined-spinal epidural);
5. The patient agrees to receive an adductor canal block;
6. American Society of Anesthesiologists class 1-3.

Exclusion Criteria:

1. Subject is < 18 years of age or >80 years of age;
2. Subject is non-English speaking;
3. Subject is known or believed to be pregnant;
4. Subject is a prisoner;
5. Subject has impaired decision-making capacity per discretion of the Investigator;
6. Symptomatic untreated gastroesophageal reflux or otherwise at risk for perioperative aspiration;
7. Any condition for which the primary anesthesia care team deems neuraxial anesthesia inappropriate;
8. Significant pre-existing neuropathy on the operative limb;
9. Significant renal, cardiac or hepatic disease per discretion of the investigator;
10. American Society of Anesthesiologists class 4-5;
11. Known hypersensitivity and/or allergies to local anesthetics;
12. Chronic Opioid Use (daily or almost daily use of opioids for > 3 months).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2018-07-16 (Actual); Study Completion 2018-07-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The American Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study aimed to obtain 70 patients to account for dropout, however was sufficiently powered if 60 patients enrolled. Study was terminated after 64th patient due to surgeon preferences.
Period: Overall Study
Arm/Group | Liposomal Bupivacaine Group | Standard Bupivacaine Group
Started | 32 | 32
Completed | 31 | 32
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine Group | Standard Bupivacaine Group | Total
Number analyzed (Participants) | 31 | 32 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (9.5) | 64.8 (6.9) | 65.8 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 21 | 46
  Male | 6 | 11 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 31 | 32 | 63

OUTCOME MEASURES:

1. Primary Outcome: 10 Meter Walk Test
Description: Time to comfortably walk 10 meters as deemed safe by physical therapy
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Liposomal Bupivacaine Group | Standard Bupivacaine Group
Number analyzed (Participants) | 31 | 32
seconds | 17.1 (8.9) | 13.4 (5.2)

2. Secondary Outcome: Pain Scores
Description: Visual Analog Scores on a scale of 1-10, where 1 is pain free and 10 is the most pain.
Time Frame: Day 0, Day 1, Day 2, Day 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liposomal Bupivacaine Group | Standard Bupivacaine Group
Number analyzed (Participants) | 31 | 32
score on a scale
  Day 0 | 4.9 (2.4) | 5.7 (2.2)
  Day 1 | 4.1 (2.3) | 4.5 (2.4)
  Day 2 | 4.4 (2.0) | 5.9 (2.6)
  Day 3 | 4.5 (2.2) | 5 (2.3)

3. Secondary Outcome: Opioid Consumption in Morphine Equivalents
Description: Total opioid consumption will be measured in all patients over the course of 3 days and converted to oral morphine equivalents so that it can be statistically compared.
Time Frame: Day 0 (OR), Day 0 (PACU), Day 1, Day 2, Day 3
Measure: Mean (Standard Deviation); unit: Morphine equivalents
Arm/Group | Liposomal Bupivacaine Group | Standard Bupivacaine Group
Number analyzed (Participants) | 31 | 32
Morphine equivalents
  Day 0 (OR) | 2.3 (6.9) | 0.5 (2.7)
  Day 0 (PACU) | 7.1 (8.4) | 5.9 (11.4)
  Day 1 | 51.2 (29.2) | 66.1 (36.0)
  Day 2 | 39.5 (28.6) | 54.8 (37.9)
  Day 3 | 25.8 (33.0) | 28.2 (20.4)

4. Secondary Outcome: Number of Participants Who Experienced Nausea
Description: Post operative nausea and vomiting as documented in the PACU and volunteered in an over the phone interview
Time Frame: Day 0, Day 1, Day 2, Day 3
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine Group | Standard Bupivacaine Group
Number analyzed (Participants) | 31 | 32
Participants
  Day 0 (PACU) | 1 | 0
  Day 1 | 12 | 11
  Day 2 | 3 | 6
  Day 3 | 4 | 6

5. Secondary Outcome: Quadriceps Strength
Description: Quadriceps Strength is measured in pounds of force using the kiio device, reported as the highest value of 3 collected.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Pounds of Force
Arm/Group | Liposomal Bupivacaine Group | Standard Bupivacaine Group
Number analyzed (Participants) | 31 | 32
Pounds of Force | 16.5 (11) | 19.2 (12.8)

ADVERSE EVENTS:
Time Frame: Up to 72 hours
Description: Any events that were deemed to be reportable events were discussed with the IRB
Arm/Group | Liposomal Bupivacaine Group | Standard Bupivacaine Group
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/32
Other Adverse Events (participants affected / at risk) | 1/31 | 0/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liposomal Bupivacaine Group (N=31) | Standard Bupivacaine Group (N=32)
Falls (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Fall as a result of prolonged quadriceps weakness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-07): https://cdn.clinicaltrials.gov/large-docs/33/NCT03182933/Prot_SAP_000.pdf